CLINICAL TRIAL: NCT03852810
Title: Patient Reported Outcomes for XEN Gel Stent Versus Trabeculectomy for the Treatment of Glaucoma
Brief Title: Satisfaction With XEN Gel Stent Versus Trabeculectomy for the Treatment of Glaucoma
Acronym: XENPRO
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: P-2016-6380
Record Dates: First submitted 2019-01-30; First posted 2019-02-25 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Receiving surgical intervention via XEN Gel Stent (XEN): Patient Reported Outcomes (PRO) will be collected before and after this particular procedure
- Receiving surgical intervention via trabeculectomy: Patient Reported Outcomes (PRO) will be collected before and after this particular procedure

SUMMARY:
This is a prospective, observational, non-interventional study of patients scheduled to receive surgical intervention either via XEN or trabeculectomy for open-angle glaucoma. The decision to treat patients with a particular surgical procedure will not be influenced by the study as the treatment decision will continue to be made by the patient and the clinician. There will be no study mandated visits or treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with OAG (Open Angle Glaucoma) and using at least 2 topical IOP-lowering medication classes in the study eye
* Scheduled to receive surgical treatment with either XEN (Xen gel stent) or trabeculectomy in the study eye
* Access to an electronic device with internet capabilities and an email address for completion of PROs (Patient Reported Outcomes)
* Be willing and able to complete PROs (Patient Reported Outcomes) at the specified time points
* Able to provide voluntary, informed consent to participate in this study

Exclusion Criteria:

* Diagnosed with angle closure glaucoma in the study eye
* Presence of a secondary glaucoma, pseudoexfoliation glaucoma, or pigmentary glaucoma
* Presence of neovascular, uveitic, or angle recession glaucoma or any glaucoma associate with vascular disorders
* Prior incisional glaucoma surgery, canal-based surgery, suprachoroidal space-based surgery (trabeculectomy, viscocanalostomy, canaloplasty, shunts of any type, collagen implants, etc.) or a cilio-ablative procedure
* Clinically significant inflammation or infection in the study eye within 30 days prior to the baseline visit (e.g. blepharitis, conjunctivitis, keratitis, uveitis, herpes simplex infection)
* History of corneal surgery, corneal opacities, or corneal disease
* Prior intraocular surgery in either eye ≤ 3 months prior to study enrollment with the exception of uncomplicated cataract surgery in either eye ≥ 1 month prior to study enrollment
* Anticipated ocular surgery in either eye within 6 months of baseline
* Concomitant cataract surgery scheduled at the time of glaucoma procedure

The study eye is defined as the eye receiving surgical intervention with either XEN or trabeculectomy.

Patients who have received prior laser trabeculoplasty will be permitted to participate if all other inclusion/exclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, approximately 150 eligible patients (75/group) will be enrolled in Canada, the UK, Germany, and Austria.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the visual function and local eye symptoms in patients receiving surgical intervention via XEN (Xen gel stent) or trabeculectomy. | 3 Months
  Visual function and local eye symptoms using the Glaucoma Symptom and Health Problem Chart (SHPC-18)
  SHPC-18 is an eighteen question survey to assess local eye and visual function symptoms caused by glaucoma or its treatments. The tool is comprised of 7 questions related to local eye symptoms, and 11 related to visual function problems. The 2-domain tool is a psychometrically validated measure of patient-reported, glaucoma-related symptoms that is responsive to treatment and discriminates the severity of glaucoma to better understand the influence of glaucoma symptoms on patients' daily life.

SECONDARY OUTCOMES:
To evaluate and compare the treatment satisfaction and expectations in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
  Patients treatment satisfaction and expectations will be measured using a study specific Glaucoma Surgery Satisfaction Survey.
To evaluate and compare work productivity in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
  Work productivity using the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem v2.0 (WPAI:SHP)
  The WPAI is a six question survey to quantitatively assess the amount of absenteeism, presenteeism, and daily activity impairment attributable to specific health problems. Participants will be asked about their employment status, the amount of hours they have missed due to their health problems, the amount of hours they have missed due to non-health problems, how many hours they worked, how much their health problems affected work productivity, and how much their health problems affected their regular daily activities for the recall period of one week
To evaluate and compare the visual acuity recovery time in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
  Visual acuity will be recorded from the patient chart and converted from the site-specific metric to EDTRS letter equivalents
To evaluate and compare the refractive change from baseline in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
To evaluate and compare the IOP (Intraocular Pressure) change from baseline in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
To evaluate and compare new onset ocular hypotensive medication use in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
To present glaucoma procedure-related adverse events in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
To evaluate glaucoma related healthcare resource utilization (HRU) by the mean number of physician office visits | 3 Months
To present post-operative medical management in patients receiving surgical intervention via XEN and trabeculectomy. | 3 Months
To evaluate glaucoma related healthcare resource utilization (HRU) by medication use | 3 Months
To present post-operative surgical management in patients receiving surgical intervention via XEN and trabeculectomy | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Campbell, Ph.D, Study Director — Allergan
Locations (10):
- Canada (4):
  - Dalhousie University, Halifax, Nova Scotia
  - Galen Eye Center, Kingston, Ontario
  - Prism Eye Institute, Mississauga, Ontario
  - Toronto Ophthalmic Research Innovation Centre, Inc, Toronto, Ontario
- Germany (3):
  - Universitat Augenklinik, Mainz
  - Ludwig-Maximilians-Universität München, Munich
  - University of Tübingen, Tübingen
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - Royal Surrey County Hospital, Guildford
  - Southend University Hospital, Southend-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
URL: http://www.allerganclinicaltrials.com/

REFERENCES:
- See also: To be considered as a site for current and future Allergan Clinical Trials, please register using the Investigator Databank link. — http://www.investigatordatabank.org/
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance — http://www.AllerganClinicalTrials.com